CLINICAL TRIAL: NCT07321093
Title: A Double-blind, Randomized Clinical Study of the Efficacy and Safety of BCD-281 in Patients With Relapsing-Remitting Multiple Sclerosis
Brief Title: A Study of the Efficacy and Safety of BCD-281 in Patients With Relapsing-Remitting Multiple Sclerosis
Acronym: MUSCAT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BCD-281-2/MUSCAT
Record Dates: First submitted 2025-11-17; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Relapsing-remitting Multiple Sclerosis (RRMS)
Keywords: Multiple Sclerosis; anti CD20; monoclonal antibody
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — ocrelizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCD-281 (Experimental): Subjects will receive 300 mg (for the first two infusions) and 600 mg via subsequent infusions.
  Interventions: Biological: BCD-281
- Ocrelizumab (Active Comparator): Subjects will receive 300 mg (for the first two infusions) and 600 mg via subsequent infusions.
  Interventions: Biological: Ocrelizumab

INTERVENTIONS:
Biological: BCD-281 — anti-CD20 monoclonal antibody
  Arms: BCD-281
Biological: Ocrelizumab — anti-CD20 monoclonal antibody
  Arms: Ocrelizumab

SUMMARY:
The aim of this study is to compare the efficacy, safety profile, pharmacokinetics, pharmacodynamics, and immunogenicity of BCD-281 and the reference drug in subjects with relapsing multiple sclerosis.

DETAILED DESCRIPTION:
The study includes the following periods:

* Screening (not more than 28 days from the date of signing the ICF).
* Double-blind period - Week 0-72.
* Open-label period - Weeks 72-96.
* Follow-up period - Weeks 96-100. The screening examination is aimed at confirming the eligibility of the subjects for the study. After confirming the eligibility, the subject will be randomized with equal probability into one of two groups (BCD-281 and the reference drug).

ELIGIBILITY:
Inclusion Criteria:

* Provided written ICF to participate in the study.
* Male and female subjects aged 18 to 55 years inclusive at the time of signing the ICF.
* Diagnosis of multiple sclerosis, established in accordance with the McDonald criteria for the diagnosis of multiple sclerosis (2017 revision).
* Relapsing-remitting multiple sclerosis.
* The total EDSS score 0-5.5 inclusive.
* Documentary evidence of the following at the time of signing the ICF:

  1. at least one relapse within the last12 months, and/or
  2. 2 relapses within the last 24 months, and/or
  3. at least 1 T1 Gd+ lesion detected on brain MRI and 1 relapse within 24 months prior to signing the ICF.
* Presence of IgG antibodies to the Varicella-Zoster virus.
* Neurological stability for 30 days prior to signing the ICF.
* Subject's willingness to discontinue previously prescribed DMTs from the day of the first administration of the IP and throughout the study.
* The ability of the subject to follow the Protocol procedures, according to the Investigator.
* Willingness of subjects of both sexes and their sexual partners of childbearing potential to use reliable methods of contraception from the time of signing ICF, throughout the study and for 5 months after the last dose of the drug in this study.

Exclusion Criteria:

* Primary progressive or secondary progressive MS.
* MS duration of more than 10 years with EDSS score of ≤2.0 at screening.
* Malignant form of MS.
* Other medical conditions that can affect the assessment of clinical picture of the MS.
* Inability to obtain high-quality MRI images and/or the presence of contraindications to MRI and the administration of gadolinium-containing contrast agents.
* Any comorbidities requiring treatment with systemic glucocorticoids and/or immunosuppressive drugs for the duration of the study, with the exception of MS.
* History of progressive multifocal leukoencephalopathy.
* Any acute or exacerbated chronic infections detected during screening that may have a negative impact on subject's safety during the study therapy.
* Concomitant diseases and/or conditions that may affect the assessment of the clinical picture of the underlying disease and/or significantly increase the risk of AEs during the study.
* Known alcohol or drug addiction, or current signs of alcohol/drug addiction.
* History of severe depression and/or a Beck Depression Inventory score of ≥16 at screening examination.
* History of a malignant disease within 5 years prior to screening.
* A diagnosis of HIV infection, hepatitis B or C .
* Inability to provide the subject with venous access.
* Pregnancy or breastfeeding, pregnancy planning and oocyte donation throughout the study and for 5 months after the last dose of ocrelizumab.
* A history of severe allergic or anaphylactic reactions to humanized and/or murine monoclonal antibodies.
* A history of using any prohibited medications or treatments defined in the study protocol.
* Abnormal laboratory blood values, as specified in the study protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 292 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Total number of T1 gadolinium-enhancing (Gd+) lesions up to Week 24. | up to Week 24
  The total number of T1 Gd+ lesions for all participants in the treatment group was calculated as the sum of the individual number of lesions at Weeks 12, 16, 20 and 24.

SECONDARY OUTCOMES:
Annualized relapse rate (ARR). | up to Week 100
  ARR was protocol-defined and calculated as the total number of relapses for all participants in the treatment group divided by the total participant-years of exposure to that treatment.
Time to first relapse. | up to Week 100
Proportion of subjects without confirmed relapses. | up to Week 100
Total number of T1 Gd+ lesions at Weeks 48, 72, 100. | up to Week 100
Total number of new or enlarged T2 lesions. | up to Week 100
Proportion of subjects without contrast-enhancing lesions. | up to Week 100
Proportion of subjects without new or enlarged T2 lesions. | up to Week 100
Total number of new hypointense T1 lesions. | up to Week 100
Change in the volume of hypointense T1 lesions. | up to Week 100
Change in the volume of T2 lesions. | up to Week 100
Combined unique active (CUA). | up to Week 100
  The total number of new T1 Gd+ lesions and new or enlarging T2 lesions, without double counting
Changes over time in the neurologic deficit according to the Expanded Disability Status Scale (EDSS). | up to Week 100
  Changes in the neurologic deficit according to EEDSS to measure disability and disease progression (from 0 to 10). An increase in the EDSS score signifies worsening disability.
Changes over time in Timed 25-Foot (7.62 meters) Walk Test performance. | up to Week 100
Changes over time in 9-Hole Peg Test (9HPT) performance. | up to Week 100
Changes over time in Symbol Digit Modalities Test (SDMT) performance. | up to Week 100
Change in quality of life using SF-36 questionnaire (36-Item Short Form Health Survey) | up to Week 100
  Change in the quality of life parameters using a SF-36 questionnaire. SF-36 (Short Form-36) questionnaire includes a total of 36 questions. Higher scores (0-100) mean better health.
Change in quality of life using EQ-5D questionnaire (EuroQol Five Dimensions) | up to Week 100
  A positive change in the Index score or a higher score generally means improvement in health.
  A negative change in the Index or a lower score means deterioration.
Proportion of subjects with confirmed disability progression (CDP). | up to Week 100
Proportion of subjects with confirmed disability worsening (CDW). | up to Week 100
The proportion of subjects with confirmed overall disability worsening. | up to Week 100
Proportion of patients with adverse reactions | up to Week 100
Proportion of patients with serious adverse reactions | up to Week 100
AUC 168-336. | up to Week 100
  Area under the drug concentration-time curve for the time interval from the measurable concentration on Day 169 to the measurable concentration on Day 337 (before the fourth administration of the investigational products).
Cmax. | up to Week 100
  Maximum observed drug concentration.
Tmax. | up to Week 100
  Time to maximum plasma concentration.
T1/2. | up to Week 100
  Terminal Elimination Half-life (T1/2) of IP.
Kel. | up to Week 100
  The elimination rate constant.
Ceoi. | up to Week 100
Ctrough. | up to Week 100
  Trough Concentration (Ctrough) of IP.
Pharmacodynamic endpoints. | up to Week 100
  PD will be evaluated based on the determination of CD19+ B-cell levels in subjects' blood.
Proportion of subjects with binding antibodies (BAbs). | up to Week 100
Proportion of subjects with neutralizing antibodies (NAbs). | up to Week 100
Time to BAb/NAb positivity. | up to Week 100

CONTACTS AND LOCATIONS:
Locations (1):
- LLC "Medis", Nizhny Novgorod, Russia

IPD SHARING:
Plan to Share IPD: No